CLINICAL TRIAL: NCT07080411
Title: A Prospective Study on the Efficacy of MR-guided Online Adaptive Radiotherapy for Locally Advanced Rectal Cancer
Brief Title: the Efficacy of MR-guided Online Adaptive Radiotherapy for Locally Advanced Rectal Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, TangYuan, Profressor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025062017264502
Record Dates: First submitted 2025-07-01; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Rectal Cancer; Adaptive Radiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRgART group (Experimental)
  Interventions: Radiation: short course radiotherapy using MR-linac

INTERVENTIONS:
Radiation: short course radiotherapy using MR-linac — Patients in the MRgART group will receive standard total neoadjuvant therapy (TNT) and surgical treatment, including short-course radiotherapy and chemotherapy, with the addition of immunotherapy at the investigator's discretion based on individual patient characteristics.

SUMMARY:
Based on preliminary findings on the motion error of the clinical target volume (CTV) in MR-guided adaptive radiotherapy (MRgART) for locally advanced rectal cancer (LARC), this study aims to reduce CTV-to-PTV margins and evaluate the complete response (CR) rate following MRgART in LARC patients. Additionally, it will investigate the safety and tolerability of MRgART, as well as its impact on:

3-year organ preservation rate

Local recurrence rate in patients under a "watch-and-wait" approach

3-year overall survival (OS), disease-free survival (DFS), and local progression-free survival (LPFS).

Furthermore, by analyzing ADC maps of the gross tumor volume (GTV), this study will characterize treatment responses and spatial deformation in metabolically active tumor subregions. These insights may inform future dose-escalation strategies for LARC radiotherapy, with the ultimate goal of improving prognosis and quality of life in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, regardless of gender;
2. Staged as II/III (cT3-T4N0 or cT2-4N+, no distant metastasis) by MRI or endoscopic ultrasound (according to the AJCC Cancer Staging Manual, 8th Edition);
3. Fibrocolonoscopy or digital rectal examination confirms the lower border of the lesion is ≤10 cm from the anal verge;
4. Pathologically confirmed or reviewed diagnosis of rectal adenocarcinoma;
5. ECOG performance status of 0-1;
6. Laboratory test results meeting the following criteria: Hemoglobin ≥ 90 g/L, white blood cells ≥ 3.5×10⁹/L; Neutrophils ≥ 1.5×10⁹/L, platelets ≥ 100×10⁹/L; Creatinine ≤ 1.0× upper normal limit (UNL), blood urea nitrogen (BUN) ≤ 1.0× UNL; Alanine aminotransferase (ALT) ≤ 1.5× UNL; Aspartate aminotransferase (AST) ≤ 1.5× UNL; Alkaline phosphatase (ALP) ≤ 1.5× UNL; Total bilirubin (TBIL) ≤ 1.5× UNL; Urine protein (-); normal bleeding and clotting time.
7. No history of allergy to 5-Fu drugs or platinum-based drugs;
8. Primary rectal cancer patients must not have undergone surgery (except palliative colostomy), chemotherapy, or other antitumor treatments from diagnosis to enrollment;
9. No prior radiation therapy to the intended treatment site;
10. Signed informed consent form.

Exclusion Criteria:

1. Presence of MRI-incompatible metal implants or claustrophobia;
2. Previous treatment with anti-PD-1/L1, anti-CTLA-4 immunotherapy, or other experimental immunotherapeutic drugs;
3. History of severe autoimmune diseases, including active inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis (e.g., Wegener's granulomatosis), etc.;
4. Symptomatic interstitial lung disease or active infectious/non-infectious pneumonia;
5. Risk factors for intestinal perforation, such as active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal malignancies, or other known predisposing conditions;
6. History of other malignancies, except for curable non-melanoma skin cancer or cervical carcinoma in situ;
7. Active infections, heart failure, myocardial infarction within the past 6 months, unstable angina, or unstable arrhythmia;
8. Physical examination or clinical findings that, in the investigator's judgment, may interfere with results or increase the patient's risk of treatment complications, or other uncontrolled medical conditions;
9. Women who are pregnant or breastfeeding;
10. Congenital or acquired immunodeficiency disorders, including human immunodeficiency virus (HIV) infection, or history of organ transplantation or allogeneic stem cell transplantation.
11. Active hepatitis B virus (HBV) infection (HBV-DNA ≥2000 U/mL), hepatitis C virus (HCV) infection, or active tuberculosis infection;
12. Prior administration of a cancer vaccine or receipt of any other vaccine within 4 weeks before treatment initiation.

    (Note: Inactivated vaccines, such as seasonal flu shots, are permitted, whereas live attenuated vaccines, such as intranasal formulations, are prohibited.)
13. Concurrent use of other immunomodulators, chemotherapy, investigational drugs, or long-term corticosteroid therapy will exclude the patient from enrollment.
14. Patients with psychiatric disorders, substance abuse, or social issues that may compromise compliance, as assessed by the investigator, will be excluded.
15. Patients with a known allergy or contraindication to the study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) | 8 weeks post chemoradiotherapy
  Absence of residual cancer cells on the final analysis of the tumor and lymph node

SECONDARY OUTCOMES:
adverse events (AE) | 2 years after radiotherapy
  Toxicity including anorexia, nausea, vomiting, diarrhoea, dermatitis, proctitis, urinary frequency/urgency according to CTCAE criteria v5.0
organ preservation rate | 8 weeks after chemoradiotherapy
  Sphincter Preservation rates 8 weeks post chemoradiotherapy at surgery.Percentage of patients who underwent sphincter salvage surgery after chemoradiotherapy
local recurrence rate (LCR) | From the completion of total neoadjuvant therapy (TNT) or post-surgery until 3 years post-treatment follow-up
disease-free survival (DFS) | From the completion of total neoadjuvant therapy (TNT) or post-surgery until 3 years post-treatment follow-up
  Time from study entry to disease recurrence or death
overall survival (OS) | From enrollment until 3 years post-treatment follow-up
  Time from study entry to death
local progression-free survival (LPFS) | From the completion of total neoadjuvant therapy (TNT) or post-surgery until 3 years post-treatment follow-up
  Time from study entry to local recurrence